CLINICAL TRIAL: NCT03232970
Title: Full Plate Diet Clinical Trial
Brief Title: Full Plate Diet Study
Acronym: FPDCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Ardmore Institute of Health (Other)
Responsible Party: Principal Investigator, Hildemar Dos Santos, MD, DrPH, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5170138
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Diet Modification

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPD group (Experimental): This group will undergo three months of weekly lectures to incorporate more fiber in their diet.
  Interventions: Other: Full Plate Diet
- FPD Control group (No Intervention): This group will receive all the assessments before, during and after the three months program period but will not attend the weekly lectures.

INTERVENTIONS:
Other: Full Plate Diet — 12 weekly sessions on how to incorporate more fiber in the diet.
  Arms: FPD group

SUMMARY:
Comparison between two groups, experimental and control. Experimental will undergo lectures on a diet to increase fiber consumption. Blood tests and anthropometric measures will be done before and after the 3-months long program. Comparisons will be made pre and post and with groups.

DETAILED DESCRIPTION:
The Full Plate Diet Clinical Trial is a study that will verify if the three months course is sufficient to change diet behavior of the participants. Forty participants will be recruited and then randomly assigned to one of two groups (20 in each group): The Experimental group will attend one weekly session with instructions on how to increase fiber intake; Control group will not have the intervention. The goal of the study is to see if the Full Plate Diet program will improve blood measures of metabolic diseases and weight.

ELIGIBILITY:
Inclusion Criteria:

* Any gender and age between 21-65 years

Exclusion Criteria:

* BMI between 25 to 35,
* no debilitating disease,
* no previous participation in the FPD program,
* no allergies to beans

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 3 months
  weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Body Fat | 3 months
  Body Fat % measured by InBody 520 BIA machine
Lipids | 3 months
  Measure of Total Cholesterol, HDL Cholesterol, LDL Cholesterol, and Triglycerides
HbA1C | 3 months
  Glycated Hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SJ, de Souza RJ, Choo VL, Ha V, Cozma AI, Chiavaroli L, Mirrahimi A, Blanco Mejia S, Di Buono M, Bernstein AM, Leiter LA, Kris-Etherton PM, Vuksan V, Beyene J, Kendall CW, Jenkins DJ, Sievenpiper JL. Effects of dietary pulse consumption on body weight: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2016 May;103(5):1213-23. doi: 10.3945/ajcn.115.124677. Epub 2016 Mar 30. PMID 27030531